Official Title of the study: Effect of Food Insulin Index on

Metabolic Parameters in Obese Adolescents

NCT number: NCT ID not yet assigned

Document Date: 2 October 2015 (The date on which the

uploaded document was approved by a human subjects

protection review board.)

This study was supported by the Scientific and Technological

Research Council of Turkey with a project number of 116S069.

# 1. Background

Obesity is one of the major public health problems in the world, and adolescence is a critical period in the development of obesity [1]. Adolescent obesity has been shown to reduce health-related quality of life and to be associated with a range of health related problems, including pre- and type 2 diabetes [1,2]. It is also well known that the high body mass index seen during the adolescence tracks substantially to adulthood [1]. Therefore, treatment of obesity in the adolescence is important in terms of both protecting the existing health and preventing the diseases in the adulthood. However, little is known about the optimal dietary approach for weight loss in obese adolescents, particularly those at risk of developing type 2 diabetes. The traditional treatment approach focuses on reducing energy intake by decreasing fat and increasing carbohydrates, but this option may not be appropriate to treat obese adolescents with insulin resistance (IR). It is speculated that this diet may lead to higher levels of postprandial glycemia and/or insulinemia and may increase IR, a potential role in the development of type 2 diabetes [2]. Furthermore, restrictive dieting may be problematic during growth and development. Thus, dietary interventions that modulate appetite and food consumption may offer alternative approaches for reducing energy intake [3].

In individuals at risk of developing type 2 diabetes, diets leading to excessive insulin secretion may increase oxidative stress and accelerate the progression of beta-cell failure [4]. Carbohydrates are the major stimulus for insulin secretion, and the glycemic index (GI) is a concept to provide the most accurate prediction of likely insulin response after consuming carbohydrate-containing foods. Recently, the role of carbohydrate quality as assessed by GI in obesity management especially for individuals with a compensatory increased insülin secretion has received considerable attention [1,2]. High-GI foods may lead to impaired balance between hormones acting in appetite stimulation (such as ghrelin) and suppression (such as incretins), thus resulting in reduced satiety and obesity. Moreover, high-GI diets, due to the rapid blood glucose and insulin response following consumption, may stimulate reduced satiety and increase voluntary energy intake [1]. Additionally, the rapid increase in postprandial plasma insülin is presumed to result in chronic stimulation of the hunger accompanied by hyperinsulinemia and lipogenesis [5]. Although carbohydrates are the major stimulus for insulin secretion, it is not the only one. Dietary proteins and fats also elicit a significant insulin response, and when combined with carbohydrates, they play a synergistic role in increasing insulin levels and reducing glycemia [2,4]. The new concept of the food insulin index (FII) allows for the testing of foods with low or no carbohydrate content, since the measure of comparison is energy as opposed to carbohydrates for the GI. For the calculation, the observed insulinemic response (area under the curve, AUC) to consumption of a 1000 kJ (239 kcal) portion of the test food divided by the insulinemic response after ingestion of a 1000 kJ portion of the reference food (either glucose or white bread) [4]. The FII concept, which directly quantifies the postprandial insulin response to a test food in comparison with an isoenergetic portion of a reference food, has been suggested to be more suitable than GI in evaluating conditions related to insulin exposure, such as obesity [6].

Nevertheless, few studies have been conducted to elucidate the role of FII in obesity. In a study investigating the effect of dietary GI and FII on body composition, it was demonstrated that a

higher dietary FII during puberty (9-14 years for girls and 10-15 years for boys) was associated with a higher percentage of body fat in young adulthood (18-25 years), although dietary GI during puberty was not related to body composition in young adulthood [7]. That study suggests a prospective adverse influence of increased insulinemia rather than increased glycemia on body composition [7]. Furthermore, a recent study has shown that diets with low insulin demand may reduce energy intake and may hence assist with weight loss in obese adolescents with IR [2]. However, the effect of FII on short-term hunger, satiety or voluntary energy intake has yet to be seen. On the other hand, single food studies found the FII as a better predictor of observed insulin responses than the carbohydrate content or GI. However, it has been yet unknown whether the FII in the context of realistic mixed meals can affect the postprandial glucose and insulin responses in obese adolescents with IR.

## 2. Objective

The aim of this study was to determine whether the FII could affect postprandial metabolic responses and appetite sensations in obese adolescents with IR, consuming two different test meals that had similar macronutrient content and GI but a 2-fold difference in FII.

#### 3. Materials and methods

## 3.1. Study design

This was a randomized, single-blind, crossover clinical trial conducted on 2 separate days, with a 1-week washout period between each study day [8]. All participants were randomly submitted to two different test meals with the following similar glycemic index (GI) and different food insulin index (FII) amounts: a low GI and low FII (LGI-LII) content, and a low GI and high FII content (LGI-HII). The order of the test meals was determined by using a computer-generated randomization sequence before recruitment. Test meals were served as a breakfast after 12-hours fasting and participants were asked to consume the meal in full, within 15 min. Venous blood samples were collected just before breakfast (t=0 min) and at time points 15, 30, 45, 60, 90, 120, 180 and 240 min after the meal [9]. Visual analogue scale (VAS) ratings were measured at the same time points, and 4 h after the breakfast, an *ad libitum* buffet-style lunch was served to each participant [10]. The primary outcomes were postprandial responses of serum glucose, insulin and C-peptide. Subjective appetite assessment were the secondary outcomes. The study design was summarized in Figure 1.

This study was conducted according to the guidelines laid down in the Declaration of Helsinki. The Clinical Research Ethics Committee of the Erciyes University approved the protocol (2015/451) on 2 October 2015, and all participants gave written informed consent.

## 3.2. Participants

Twenty two obese adolescents with IR who attended the outpatient clinic of the Pediatric Endocrinology, at the Child Hospital of Erciyes University, Kayseri, Turkey were selected on the basis of the following criteria: aged 12-18 years, age- and sex-specific body mass index (BMI) ≥95th percentile of the growth-reference data, new diagnosis and not receiving any treatment, and HOMA-IR >3.16. Exclusion criteria included hypertension, cardiovascular

disease, diabetes mellitus or any other significant metabolic, endocrine or gastrointestinal disease, use of tobacco or alcohol, taking any medications, and having difficulties for physical activity.

#### 3.3. Clinical evaluation

All participants underwent a detailed physical examination by the pediatric endocrinologist before included in the study. Obesity was defined according to the BMI (weight in kg/height in m²) ≥95th percentile of the WHO 2007 growth-reference for 5-19 years [11,12]. IR was assessed through Homeostatic Model Assessment for IR (HOMA-IR) which is a valid tool for evaluating IR in children and adolescents [13]. This index was calculated as follows: HOMA-IR = [fasting insulin level (µU/mL) × fasting glucose level (mmol/L)] / 22.5 [14]. HOMA-IR>3.16 was used as a threshold for IR [15]. Furthermore, pubertal maturation was determined using Tanner-Marshall descriptive standards by the pediatric endocrinologist [16,17]. Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured by aneroid sphygmomanometer in the sitting position after 10 min of rest [18].

## 3.4.Anthropometric measurements

Body height and weight were measured using an automatic height gauge scale (DENSI GL150, Istanbul, Turkey) sensitive to 10-200 kg±50 g and 90-200 cm±1 mm. The measurements were made with the participants in the minimum clothing possible, without shoes, standing barefoot, keeping shoulders in a relaxed position, arms hanging freely and head in the Frankfort horizontal plane [19]. Waist, hip and neck circumference were measured to the nearest 0.1 cm using a non-elastic tape with the participants standing, with the face directed towards, shoulders relaxed, and the tape was positioned at a level parallel to the floor. Waist circumference was measured at the end of normal expiration and the measurement site was midway between the lowest rib and the top of the iliac crest. Hip circumference was measured at the widest part of the hip at the level of the greater trochanter [19]. Neck circumference was measured with the their head held erect, eyes facing forward and the neck in a horizontal plane at the level of the most prominent portion of the thyroid cartilage [20]. All measurements were done in duplicate for each participant. If the two measurements differed by more than 1%, a third measurement was taken. All three measurements were recorded and the mean of the two nearest measures was calculated [21]. BMI was calculated as weight (kg) divided by the square of height (m<sup>2</sup>) [19], and converted age- and sex-specific z-score according to WHO criteria [12].

Body fatness was estimated by the bio-electrical impedance analysis method, by a segmental body composition analyser (BCA), Tanita BC-418MA (Tanita Corporation, Tokyo, Japan) [22]. Before the analysis, participants were asked to refrain from food or drink in the four hours prior to measurement, and to wear light clothes [19]. Participants stood with bare feet over the analyzer holding handgrips in each hand. The segmental BCA shows separate body mass readings for body fat (BF, kg), trunk fat (TF, kg), fat free mass (FFM, kg) and muscle mass (MM, kg). Also, body water (BW, kg) and basal metabolic rate (BMR, kcal) was determined by the BCA.



**Figure 1.** The study design

## 3.5.Dietary and physical activity assessment

Participants' dietary intakes were assessed by the 24-hours dietary recalls using a photographic atlas of food portion sizes to quantify the data in the beginning of study and on the day of each meal test [8,23]. Diet composition was analyzed by the BeBiS Nutrition Information System software version 7.2 [24]. This database contains Turkish food composition tables for all foods.

Physical activity level was evaluated by the IPAQ short form, a validated survey instrument [25]. The 7-item IPAQ records self-reported physical activity in the last seven days [26]. Responses were converted to Metabolic Equivalent Task (MET) minutes per week according to the IPAQ scoring protocol [26].

At the first visit, clinical, nutritional and physical activity evaluations were performed. Visits 2 and 3 were the test days. Participants received each test meal in a randomly assigned order on two different mornings separated by a washout period of 1-week when they were asked to maintain their usual diet and physical activity [27]. On the day before each test meal, participants were instructed to eat a standard evening meal at 20:00 h and to refrain from eating and/or drinking (except for water) and/or doing any physical activity beyond that of their typical daily activities [28]. Moreover, female participants were tested within the follicular phase of their menstrual cycle (3–10 d after onset of menses) to avoid any effect of menstrual cycle phase on appetite [29-31].

On the each testing day, participants arrived in the testing room at 08.00 h following a 12-h fast and were asked by the dietitian to record their 24-h food and beverage consumption. Participants' body weight, height, body composition and baseline appetite were measured before eating the test meal [8]. Also, a catheter was introduced in an antecubital vein by a registered nurse and a first blood sample was immediately drawn for baseline measurements (time zero) [32]. At 08:30 h participants received the test meal blinded to its nutritional characteristics and were asked to consume within 15 min [9,33]. During the postprandial period, participants remained at rest in the testing room and blood samples were obtained at time points 15, 30, 45, 60, 90, 120, 180, and 240 min [9]. Appetite scale was applied at the same time points [10]. Moreover, participants were asked to assess the organoleptic characteristics (visual appeal, smell, taste, aftertaste and palatability) of test meal by VAS at 15 min (immediately after consuming test meal) [34]. No food or drink other than water was allowed following consumption of the test meal until the ad libitum lunch. Water was available ad libitum throughout the first trial; however, the volume consumed was measured and the participants drank the same volume during the second trial [35,36]. Participants were permitted to watch movies, read, or play with electronic devices (laptop computer, mobile phone etc.) or undertake other similar sedentary activities throughout each study day but were not allowed to sleep [10,28,37].

At 240 min after the test breakfast, participants were presented with an *ad libitum* lunch following blood sample collection and appetite sensation measurement [28,38]. Participants selected from a buffet-style meal consisting of a variety of foods from each food group (meatballs, chicken nuggets, pasta with tomato sauce, potatoes salad, carrots salad, yoghurt, white bread, grain bread, cookies, apple, mandarin and banana) [27,28,39] with bottled water and some fruit juices (black cherry juice and peach juice) as a beverage [29,40]. These foods were determined according to their preference for adolescents to consume, frequent consumption in the Central Anatolia region, and be widely preferred in similar studies. During the lunch, participants were left alone in a quiet room with controlled lightning and ambient room temperature, and asked to consume whatever they wanted and to eat until they felt comfortably full [28,38]. Foods were weighted or measured to the nearest 0.1 g before consumption, and any remaining food was reweighed to determine intake at lunch. Energy and macronutrient values were calculated using The National Food Composition Database (TurKomp) [41] and manufacturer labelling. Moreover, the first food to start eating, all foods

selected by participants, and duration of meal were recorded at lunchtime. All foods served at breakfast and lunch were prepared by the research dietitian in the kitchen of the Nutrition Laboratory in the Faculty of Health Sciences, Erciyes University, Kayseri, Turkey on the day of each test meal.

### 3.7.Test meals composition

Test meals were matched for macronutrients and GI but had a 2-fold difference in FII. The nutritional composition and weight of the test breakfasts was shown in Table 1.

GI and FII of foods in test meals were estimated by using the GI and FII for 1000-kJ portions of foods tables published by Bao et al. [42], with glucose as the reference food. The average meal GI and FII were calculated as follows [6]:

where n is the number of foods consumed,  $GI_a$  is the GI for food a,  $II_a$  is the II for food a,  $AvCHO_a$  is the available carbohydrate content per serving of food a,  $Energy_a$  is the energy content per serving of food a, and  $Energy_a$  is the consumption frequency of one serving of food a during the meal.

**Table 1.** Nutritional composition, GI, and FII of the component foods in test meals

| | Weight | Energy | AvCHO* | Protein | Fat | GI | FII |
|---|---|---|---|---|---|---|---|
| | <b>(g)</b> | (kJ[kcal]) | <b>(g)</b> | <b>(g)</b> | <b>(g)</b> | (%) | (%) |
| LGI-LII | | | | | | | |
| Grain bread | 25 | 217(52) | 9.6 | 2.4 | 0.4 | 50 | 41 |
| Egg (boiled) | 42 | 246(59) | 0.0 | 5.4 | 4.2 | 0 | 23 |
| Milk (full-fat) | 210 | 550(131) | 10.4 | 6.0 | 7.1 | 31 | 24 |
| Breakfast cereal | 40 | 597(143) | 23.9 | 5.4 | 2.4 | 30 | 23 |
| Apple | 200 | 469(112) | 24.9 | 0.9 | 0.9 | 36 | 43 |
| Total | | 2079(497) | 68.8 | 20.2 | 15.1 | 35 | 30 |
| LGI-HII | | | | | | | |
| Grain bread | 18 | 157(38) | 6.9 | 1.7 | 0.3 | 50 | 41 |
| Cheddar cheese | 22 | 373(89) | 0.0 | 5.6 | 7.5 | 0 | 33 |
| Yogurt (low-fat strawberry) | 350 | 1383(330) | 54.0 | 13.8 | 6.9 | 31 | 84 |
| Banana | 45 | 146(35) | 8.0 | 0.3 | 0.1 | 52 | 59 |
| Total | | 2059(492) | 68.8 | 21.4 | 14.8 | 35 | 70 |

<sup>\*</sup>AvCHO, available carbohydrate including sugars and starch, excluding fiber.

## 3.8.Laboratory measurements

Fasting blood glucose (FBG), insulin, total cholesterol (TC), high-density lipoprotein (HDL), low-density lipoprotein (LDL), triglyceride (TG), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were measured after a 12-h fast. Biochemical parameters were determined by using enzymatic kits from Roche Diagnostics with a Roche Cobas® 8000 modular analyzer series. On test days, approximately 2 mL of blood were drawn for each time points (0, 15, 30, 45, 60, 90, 120, 180 and 240 min) to determine serum glucose, insulin and Cpeptide levels. Blood samples after collecting were immediately centrifuged and assayed. Serum glucose was measured by a spectrophotometric method (Roche Cobas® 8000 Modular Analyzer Series, c701 module), and serum insulin and C-peptide by electrochemiluminescence immunoassay (ECLIA) method (Roche Cobas® 8000 Modular Analyzer Series, e602 module) using Roche kits (Roche Diagostics, Mannheim, Germany).

# 3.9. Assessment of appetite sensations

Subjective assessment of appetite sensations was performed by using a visual analogue scale (VAS) composed of lines (of 100 mm in length) with words anchored at each end, expressing the most positive and the most negative rating [34]. VAS was used to assess appetite scores (hunger, fullness, desire to eat, and prospective food consumption), desire for specific food types (sweet, salty, savoury, and fatty) and the palatability of test meals (visual appeal, smell, taste, aftertaste, and palatability). As shown in Figure 2, a series of VAS were administered using the paper-and-pen method at specific time-points (immediately before and after consuming test meal, and thereafter at 30, 45, 60, 90, 120, 180 and 240 min for 4 hours) during the examination period. Participants were asked to make a single vertical mark at the appropriate point between the 2 anchors on each scale corresponding to their feelings. A new VAS booklet was provided to participants for each rating time, and nobody could compare to his/her previous ratings when marking the VAS. Appetite scores were quantified by measuring the distance in millimeters between the left end of each line and the mark [8]. The questions on appetite, desire for specific food types and palatability of test meals, and anchored answers were as follows [34]:

- Hunger, "How hungry do you feel?" (not at all hungry as hungry as I ever felt).
- Fullness, "How full do you feel?" (not at all full totally full).
- Desire to eat, "How strong is your desire to eat?" (very weak very strong).
- Prospective food consumption, "How much do you think you can eat?" (no food at all

   a large amount of food).
- Desire for specific food types, "Would you like to eat something sweet/ salty/ savoury/ fatty?" (No, not at all Yes, very much)
- Palatability of test meals, "How is the visual appeal/ smell/ taste/ palatability of test meal?" (Good – Bad), and "Is there any perceived taste in your mouth after test meal?" (Much – None)



Figure 2. Study protocol on test days

### 4. Statistical Analysis Plan

### 4.1. Sample size and power analysis

Preliminary study was carried out to determine a sample size, and power analysis was conducted by using PASS 11 (power analysis statistical system). A power-based sample size calculation revealed that 16 participants were needed to provide 80% power to detect 5% difference between groups in areas under the curve (AUC) assessed after consumption test meals with similar GI and different FII amounts in obese adolescents with IR. It was decided to complete the study with 20 participants considering 25% losses. However, this study was concluded with 15 participants although 22 participants were recruited. Two enrolled participant declined to eat second test breakfast after consuming first test breakfast. One participant with the IPAQ score >1.2 was excluded from the study because of a decision about including only sedentary participants defined as scoring ≤1.2 on the IPAQ due to a possible effect of physical activity level on postprandial metabolic response [35]. Moreover, two participant at Tanner stage 3 or 4 were excluded due to a decision about including only participants completed pubertal maturation at Tanner stage 5 for the purpose of minimizing a possible effect of puberty on postprandial metabolic response since hormonal regulation may vary in each pubertal stages [7]. Finally, two participant were not included to the analysis of data because of hemolysis in their blood samples at some time points, leaving a total of 15 participants that were assessed for the main outcomes. When power analysis was repeated, that sample size had 81.2% power to detect differences in primary outcomes among the test meals at alpha level of 0.05.

# 4.2. Data analysis

Statistical analysis was performed using the Statistical Package for the Social Sciences (version 22.0; IBM SPSS Statistics) software. Data were expressed as the number (n) and percentage (%) for categorical variables, and means ± SDs, medians (25th–75th percentiles) for continuous variables. Normality was assessed using the histogram and normal Q-Q plots, and also Shapiro-Wilk test. Furthermore, continuous variables were examined for skewness and kurtosis, and log-transformed before analysis and reported back-transformed geometric means (G) ± standard error (S.E) when required [43]. Differences between groups were tested using t-tests. Categorical variables were compared by the chi-square tests. Wilcoxon signed rank tests were used for continuous variables without normal distributions. Postprandial responses for metabolic parameters and appetite sensations were quantified as area under the curve (AUC) calculated according to the trapezoidal rule [8,33]. As an estimate of glucose-adjusted insulin response, the index of insulin response to glucose was calculated as an insulin/glucose ratio by using serum glucose and insulin levels at time points [9]. A Student's 2-tailed t test for paired data was applied to determine statistical differences between AUCs. In addition, between-group comparisons were analyzed by using 2-factor (diet x time) repeated-measures analysis of variance (ANOVA), and Bonferroni post hoc tests were applied to significant group x time interactions. Baseline values for each variable were compared between groups by using paired t tests. In the event of a significant t statistic, baseline values were used as a covariate in the 2factor repeated-measures ANOVA. For all statistical analyses, p values less than 0.05 were considered to have statistical significance [44].

#### REFERENCES

- 1. Murakami K, McCaffrey TA, Gallagher AM, Neville CE, Boreham CA, Livingstone MB. Dietary glycemic index and glycemic load in relation to changes in body composition measures during adolescence: Northern Ireland Young Hearts Study. Int J Obes (Lond) 2014;38:252-8.
- 2. Joslowski G, Halim J, Goletzke J, et al. Dietary glycemic load, insulin load, and weight loss in obese, insulin resistant adolescents: RESIST study. Clin Nutr 2015;34:89-94.
- 3. Liu AG, Puyau RS, Han H, Johnson WD, Greenway FL, Dhurandhar NV. The effect of an egg breakfast on satiety in children and adolescents: a randomized crossover trial. Journal of the American College of Nutrition 2015;34:185-90.
- 4. Bao J, de Jong V, Atkinson F, Petocz P, Brand-Miller JC. Food insulin index: Physiologic basis for predicting insulin demand evoked by composite meals. Am J Clin Nutr 2009;90:986-92.
- 5. Kong AP, Chan RS, Nelson EA, Chan JC. Role of low-glycemic index diet in management of childhood obesity. Obes Rev 2011;12:492-8.
- 6. Nimptsch K, Brand-Miller JC, Franz M, Sampson L, Willett WC, Giovannucci E. Dietary insulin index and insulin load in relation to biomarkers of glycemic control, plasma lipids, and inflammation markers. Am J Clin Nutr 2011;94:182-90.
- 7. Joslowski G, Goletzke J, Cheng G, Günther AL, Bao J, Brand-Miller JC, Buyken AE. Prospective associations of dietary insulin demand, glycemic index, and glycemic load

- during puberty with body composition in young adulthood. Int J Obes (Lond) 2012;36:1463-71.
- 8. Silva FM, Kramer CK, Crispim D, Azevedo MJ. A high-glycemic index, low-fiber breakfast affects the postprandial plasma glucose, insulin, and ghrelin responses of patients with type 2 diabetes in a randomized clinical trial. J Nutr 2015;145:736-41.
- 9. Runchey SS, Valsta LM, Schwarz Y, Wang C, Song X, Lampe JW, Neuhouser ML. Effect of low- and high-glycemic load on circulating incretins in a randomized clinical trial. Metabolism 2013;62:188-95.
- 10. Yip W, Wiessing KR, Budgett S, Poppitt SD. Using a smaller dining plate does not suppress food intake from a buffet lunch meal in overweight, unrestrained women. Appetite 2013;69:102-7.
- 11. Mirza NM, Palmer MG, Sinclair KB, McCarter R, He J, Ebbeling CB, Ludwig DS, Yanovski JA. Effects of a low glycemic load or a low-fat dietary intervention on body weight in obese Hispanic American children and adolescents: A randomized controlled trial. Am J Clin Nutr 2013;97:276-85.
- 12. <a href="http://www.who.int/growthref/who2007\_bmi\_for\_age/en/">http://www.who.int/growthref/who2007\_bmi\_for\_age/en/</a>.
- 13. Keskin M, Kurtoglu S, Kendirci M, Atabek ME, Yazici C. Homeostasis model assessment is more reliable than the fasting glucose/insulin ratio and quantitative insulin sensitivity check index for assessing insulin resistance among obese children and adolescents. Pediatrics 2005;115:e500-3.
- 14. Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia 1985;28:412-9.
- 15. Karatzi K, Moschonis G, Barouti AA, Lionis C, Chrousos GP, Manios Y; Healthy Growth Study Group. Dietary patterns and breakfast consumption in relation to insulin resistance in children: The Healthy Growth Study. Public Health Nutr 2014;17:2790-7.
- 16. Marshall WA, Tanner, J.M. . Variations in pattern of pubertal changes in girls. Arch Dis Child 1969;44:291-303.
- 17. Marshall WA, Tanner, J.M. Variations in the pattern of pubertal changes in boys. Arch Dis Child 1970;45:13-23.
- 18. Gülmez R, Demirel F, Emir S. Obez çocuk ve ergenlerde obeziteye eşlik eden endokrin ve metabolik bozukluklar ve ilişkili faktörler. Türkiye Çocuk Hast Derg 2015;2:104-12.
- 19. Pekcan G. Beslenme durumunun saptanması. In: Baysal A, Aksoy M, Besler T, Bozkurt N, Keçecioğlu S, Mercanlıgil SM, Merdol TK, Pekcan G, Yıldız E (ed). Diyet El Kitabı. Ankara: Hatiboğlu Yayınları; 2013. p. 67-142.
- 20. Nafiu OO, Burke C, Lee J, Voepel-Lewis T, Malviya S, Tremper KK. Neck circumference as a screening measure for identifying children with high body mass index. Pediatrics 2010;126:e306-10.
- 21. Van Lippevelde W, Te Velde SJ, Verloigne M, et al. Associations between family-related factors, breakfast consumption and BMI among 10- to 12-year-old European children: the cross-sectional ENERGY-study. PloS one 2013;8:e79550.
- 22. https://tarti.com/tanita-bc-418-vucut-analiz-urun35.html.
- 23. Warren JM, Henry CJ, Simonite V. Low glycemic index breakfasts and reduced food intake in preadolescent children. Pediatrics 2003;112:e414.

- 24. BeBİS (Beslenme Bilgi Sistemi) Bilgisayar Yazılım Programı Versiyon 7 (Ebispro für Windows, Stuttgart, Germany; Türkçe Versiyonu).
- 25. Saglam M, Arikan H, Savci S, et al. International physical activity questionnaire: reliability and validity of the Turkish version. Perceptual and motor skills 2010;111:278-84.
- 26. Committee IR. Guidelines for data processing and analysis of the International Physical Activity Questionnaire (IPAQ) short and long forms Retrieved September 2008; 2005.
- 27. Mehrabani S, Safavi SM, Mehrabani S, et al. Effects of low-fat milk consumption at breakfast on satiety and short-term energy intake in 10- to 12-year-old obese boys. European journal of nutrition 2015.
- 28. Baum JI, Gray M, Binns A. Breakfasts Higher in Protein Increase Postprandial Energy Expenditure, Increase Fat Oxidation, and Reduce Hunger in Overweight Children from 8 to 12 Years of Age. The Journal of nutrition 2015;145:2229-35.
- 29. Beck EJ, Tosh SM, Batterham MJ, Tapsell LC, Huang XF. Oat beta-glucan increases postprandial cholecystokinin levels, decreases insulin response and extends subjective satiety in overweight subjects. Molecular nutrition & food research 2009;53:1343-51.
- 30. Chowdhury EA, Richardson JD, Tsintzas K, Thompson D, Betts JA. Carbohydrate-rich breakfast attenuates glycaemic, insulinaemic and ghrelin response to ad libitum lunch relative to morning fasting in lean adults. The British journal of nutrition 2015;114:98-107.
- 31. Chowdhury EA, Richardson JD, Tsintzas K, Thompson D, Betts JA. Effect of extended morning fasting upon ad libitum lunch intake and associated metabolic and hormonal responses in obese adults. International journal of obesity 2015.
- 32. Bidwell AJ, Fairchild TJ, Wang L, Keslacy S, Kanaley JA. Effect of increased physical activity on fructose-induced glycemic response in healthy individuals. European journal of clinical nutrition 2014;68:1048-54.
- 33. Jakubowicz D, Wainstein J, Ahrén B, Bar-Dayan Y, Landau Z, Rabinovitz HR, Froy O. High-energy breakfast with low-energy dinner decreases overall daily hyperglycaemia in type 2 diabetic patients: A randomised clinical trial. Diabetologia 2015;58:912-9.
- 34. Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. International journal of obesity and related metabolic disorders: journal of the International Association for the Study of Obesity 2000;24:38-48.
- 35. Stevenson EJ, Astbury NM, Simpson EJ, Taylor MA, Macdonald IA. Fat oxidation during exercise and satiety during recovery are increased following a low-glycemic index breakfast in sedentary women. J Nutr 2009;139:890-7.
- 36. Zakrzewski JK, Stevenson EJ, Tolfrey K. Effect of breakfast glycemic index on metabolic responses during rest and exercise in overweight and non-overweight adolescent girls. Eur J Clin Nutr 2012;66:436-42.
- 37. Griffioen-Roose S, Mars M, Finlayson G, Blundell JE, de Graaf C. The effect of within-meal protein content and taste on subsequent food choice and satiety. Br J Nutr 2011;106:779-88.

- 38. Dalton M, Hollingworth S, Blundell J, Finlayson G. Weak Satiety Responsiveness Is a Reliable Trait Associated with Hedonic Risk Factors for Overeating among Women. Nutrients 2015;7:7421-36.
- 39. Doyon CY, Tremblay A, Rioux LE, et al. Acute effects of protein composition and fibre enrichment of yogurt consumed as snacks on appetite sensations and subsequent ad libitum energy intake in healthy men. Applied physiology, nutrition, and metabolism = Physiologie appliquee, nutrition et metabolisme 2015;40:980-9.
- 40. Aston LM, Stokes CS, Jebb SA. No effect of a diet with a reduced glycaemic index on satiety, energy intake and body weight in overweight and obese women. Int J Obes (Lond) 2008;32:160-5.
- 41. TÜBİTAK. Ulusal Gıda Kompozisyon Veri Tabanı TürKomp. Versiyon 1.0 ed: T.C. Gıda, Tarım ve Hayvancılık Bakanlığı; 2014.
- 42. Bao J, Atkinson F, Petocz P, Willett WC, Brand-Miller JC. Prediction of postprandial glycemia and insulinemia in lean, young, healthy adults: glycemic load compared with carbohydrate content alone. Am J Clin Nutr 2011;93:984-96.
- 43. Akin L, Kendirci M, Narin F, et al. The endocrine disruptor bisphenol A may play a role in the aetiopathogenesis of polycystic ovary syndrome in adolescent girls. Acta Paediatr 2015;104:e171-7.
- 44. Karagöz Y. SPSS 22 Uygulamalı Biyoistatistik. Güncellenmiş 2.Basım edition. Ankara: Nobel Yayınevi; 2015.